CLINICAL TRIAL: NCT05020340
Title: Reattempt of External Cephalic Version After Regional Anaesthesia Immediately Before a Caesarean Delivery - a Randomized Controlled Trial
Brief Title: External Cephalic Version Immediately Before a Caesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW 21-086
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Malpresentation Before Labor Affecting Fetus or Newborn
MeSH Terms: interventions — Version, Fetal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): External cephalic version
  Interventions: Procedure: External cephalic version
- Control (No Intervention): ECV will not be performed.

INTERVENTIONS:
Procedure: External cephalic version — In the intervention group, ECV will be performed by two operators with one of them having experience of ≥ 5 successful ECV. The procedure will be performed by the first operator under real time continuous ultrasonographic guidance. The fetal head and buttock will be grasped by both hands and attempt to rotate the fetus to a longitudinal lie either in a clockwise or anti-clockwise fashion. The second operator will perform the ECV if the first operator fails the procedure.
  Arms: Intervention

SUMMARY:
Fetal malpresentation at term affects around 5% of pregnancy and breech presentation is the most common type of malpresentation. It is a common indication for a Caesarean delivery. External cephalic version (ECV) refers to turning the fetus manually and aims to increase the success of vaginal birth by reducing the need for Caesarean section.

DETAILED DESCRIPTION:
Several factors affect the chance of a successful ECV which include multiparity, use of tocolytic and regional anaesthesia during the procedure. Anticipating or not tolerating a painful procedure is another factor that affects the willingness to and success of ECV.

ECV can be reattempted under regional anaesthesia immediately just before the Caesarean section to increase the vaginal birth rate in women who have failed an ECV. Therefore, the aim of this study is to evaluate whether this approach could increase the rate of vaginal birth and reduce the non-cephalic presentation at labour and Caesarean section rate.

ELIGIBILITY:
Inclusion Criteria:

* All women age ≥ 18 years old
* Singleton pregnancy
* Malpresentation
* Have failed an ECV
* Pregnant ≥ 37 weeks of gestation

Exclusion Criteria:

* Condition requiring emergency delivery
* Other indication for Caesarean section
* History of antepartum haemorrhage in the past 7 days
* Oligohydraminos with amniotic fluid index <5cm
* Intrauterine growth restriction with abnormal fetal Doppler or cardiotocography
* Rhesus isoimmunization
* Rupture of membranes
* Gross fetal anomaly
* Major uterine anomaly
* Contraindication or refusal to regional anaesthesia
* Spontaneous cephalic version on the day of scheduled Caesarean section

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Vaginal birth | Delivery
  Vaginal birth

IPD SHARING:
Plan to Share IPD: No